CLINICAL TRIAL: NCT01119027
Title: Assessing Effectiveness of Laparoscopic Colorectal Surgical Skills
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Conor Delaney, MD, PhD, Principal Investigator, University Hospitals Cleveland Medical Center
Other Study IDs: 07-09-04; 07-09-04 (Other: Unversity Hospitals Case Medical Center)
Record Dates: First submitted 2010-04-29; First posted 2010-05-07 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2012-11

CONDITIONS: Colonic Diseases
Keywords: Laparoscopic Colectomy; Colorectal Skills Training
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Surgeons: Surgeons and trainee surgeons attending laparoscopic colorectal training courses will be recruited to study using different training models to compare each model and correlate outcomes with each model to pre-course experience. .
- Trainee Surgeons: Surgeon and trainee surgeons attending laparoscopic colorectal training courses will be recruited to study using different training models to compare each model and correlate outcomes with each model to pre-course experience.

SUMMARY:
The purpose of this study is to improve the investigators understanding of different training methods in laparoscopic colon surgery.

DETAILED DESCRIPTION:
In this study the investigators use an objective evaluation system which deconstructs laparoscopic colectomy into its component steps. Critical components of the procedure as well as overall operative performance can be evaluated. This is applied to surgeons and trainee surgeons attending laparoscopic colorectal training courses using different training models to compare each model and correlate outcomes with each model to pre-course experience. This project is aimed at better educating trainers and getting better information on the validity of new training models for laparoscopic colectomy.

Aims of Project

* To observe and assess surgical technique during laparoscopic colorectal skills training courses using a previously validated tool for formal assessment of surgical technical skills.
* To evaluate technical errors and patterns of error during training at laparoscopic colectomy.
* To determine outcomes and error rates with different training models and correlate these with prior surgical experience.

Number of participants/subjects in research:

Subjects will be recruited in several sites:

* the principal investigators facility at University Hospitals of Cleveland Case Medical Center, where surgeons from outside institutions visit regularly for training courses
* Society of American Gastrointestinal and Endoscopic Surgeons (SAGES) Laparoscopic colorectal training courses, where surgeons participate in courses with invited faculty at national meetings (the PI is national Program Director and runs these courses).
* American Society of Colorectal Surgeons (ASCRS) Laparoscopic colorectal training courses, where surgeons participate in courses with invited faculty at national meetings (the PI is national Program Director and runs these courses).

Course attendees will be informed before the start of an appropriate laparoscopic course that the study is being performed. The study will be explained to them in detail and they will be given a copy of the appropriate paperwork to review. Verbal consent will be requested. It will be explained to them that they should feel under no pressure to participate in the study, and that if they do participate that these data are not used for their evaluation. The number of cases of components of cases that they perform will not be related to participation or non-participation in the trial.

Study Design This is an observational study in which trainees' technical surgical skills are evaluated while performing specific steps of laparoscopic colectomy cases, as outlined in the accompanying datasheets. The plan is to enroll 200 participants.

At the completion of each case, forms will be completed by the trainee, and by the teaching / supervising surgeon. Independent observers cannot be used, as only an attending laparoscopic colorectal surgeon is adequately skilled to score the resident performing the case, and it is not feasible to have a second attending surgeon present during each case.

Dr Delaney will score trainees when possible using the standardized form. For courses at University Hospitals Case Medical Center (UHCMC), the colorectal faculty will be instructed in standardized assessment, and will also assess trainees. For courses at SAGES or ASCRS, the course faculty will be shown the training assessments and directed in the standardized assessment prior to evaluations.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be recruited in several sites:

* The principal investigators facility at University Hospitals of Cleveland Case Medical Center, where surgeons from outside institutions visit regularly for training courses
* Society of American Gastrointestinal and Endoscopic Surgeons (SAGES) Laparoscopic colorectal training courses, where surgeons participate in courses with invited faculty at national meetings (the PI is national Program Director and runs these courses).
* American Society of Colorectal Surgeons (ASCRS) Laparoscopic colorectal training courses, where surgeons participate in courses with invited faculty at national meetings (the PI is national Program Director and runs these courses).

Exclusion Criteria:

Not applicable

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Surgeons and trainee surgeons attending laparoscopic colorectal training courses.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To observe and assess surgical technique used by surgeons and surgeon trainees in attendance during laparoscopic colorectal skills training courses. | one year
  To observe and assess surgical technique by surgeons and surgeon trainees in attendance during laparoscopic colorectal skills training courses using a previously validated tool for formal assessment of surgical technical skills.

SECONDARY OUTCOMES:
To evaluate technical errors and patterns of error by surgeons and surgeon trainees during training of laparoscopic colectomy. | one year
  To evaluate technical errors and patterns of error of surgeons and surgeon trainees during training at laparoscopic colectomy. To determine outcomes and error rates with different training models and correlate these with prior surgical experience

CONTACTS AND LOCATIONS:
Overall Officials: Conor P Delaney, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States